CLINICAL TRIAL: NCT01016691
Title: Safety and Efficacy of a Drug Delivery System in Glaucoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vistakon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR-1649
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Results first posted 2012-01-27 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-02

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- High Dose Drug Device/ bimatoprost 0.03% (Experimental): drug device containing 65 micrograms of bimatoprost released over 4 days (first period) bimatoprost 0.03% ophthalmic solution for one day (second period).
  Interventions: Drug: High Dose Drug Device; Drug: bimatoprost 0.03%
- Low Dose Drug Device / bimatoprost 0.03% (Experimental): drug device containing 45 micrograms of bimatoprost released over 4 days (first period) bimatoprost 0.03% ophthalmic solution for one day (second period).
  Interventions: Drug: Low Dose Drug Device; Drug: bimatoprost 0.03%
- Placebo Device / bimatoprost 0.03% (Other): placebo drug device worn over 4 days (first period) bimatoprost 0.03% ophthalmic solution for one day (second period).
  Interventions: Drug: Placebo Device; Drug: bimatoprost 0.03%

INTERVENTIONS:
Drug: High Dose Drug Device — device inserted for 4 days
  Arms: High Dose Drug Device/ bimatoprost 0.03%
Drug: Low Dose Drug Device — device inserted for 4 days
  Arms: Low Dose Drug Device / bimatoprost 0.03%
Drug: Placebo Device — device inserted for 4 days
  Arms: Placebo Device / bimatoprost 0.03%
Drug: bimatoprost 0.03% — one drop in each eye on one day only

SUMMARY:
Evaluation of the ocular safety and efficacy of a drug delivery system in open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman 21 years of age or greater
* Open angle glaucoma or ocular hypertension
* Corrected visual acuity in each eye of 20/200 or better

Exclusion Criteria:

* Previous glaucoma intraocular surgery or refractive surgery
* Planned contact lens use during the study
* Clinically significant ocular or systemic disease that might interfere with the study
* Use of chronic corticosteroids by any route

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2009-10; Primary Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Miami, Florida
  - Philadelphia, Pennsylvania
  - Mt. Pleasant, South Carolina
  - Rapid City, South Dakota
  - Maryville, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- High Dose Drug Device/ Bimatoprost 0.03%: high dose drug device during first period, bimatoprost 0.03% during second period.
- Low Dose Drug Device / Bimatoprost 0.03%: low-dose drug device during first period, bimatoprost 0.03% during second period.
- Placebo Device / Bimatoprost 0.03%: placebo device during first period, bimatoprost 0.03% during second period.
Period: Overall Study
Arm/Group | High Dose Drug Device/ Bimatoprost 0.03% | Low Dose Drug Device / Bimatoprost 0.03% | Placebo Device / Bimatoprost 0.03%
Started | 17 | 12 | 18
Completed | 17 | 12 | 18
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Drug Device/ Bimatoprost 0.03% | Low Dose Drug Device / Bimatoprost 0.03% | Placebo Device / Bimatoprost 0.03% | Total
Number analyzed (Participants) | 17 | 12 | 18 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (9.78) | 66.3 (11.37) | 63.1 (9.07) | 63.4 (8.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 10 | 30
  Male | 5 | 4 | 8 | 17
Region of Enrollment [Number; unit: participants]
  United States | 17 | 12 | 18 | 47

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Intraocular Pressure at Day 1
Time Frame: Baseline to Day 1
Population: per-protocol population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | High Dose Drug Device/ Bimatoprost 0.03% | Low Dose Drug Device / Bimatoprost 0.03% | Placebo Device / Bimatoprost 0.03%
Number analyzed (Participants) | 14 | 11 | 15
mmHg | -4.16 (3.409) | -4.57 (3.645) | -0.60 (2.331)

2. Secondary Outcome: Mean Change in Intraocular Pressure at Day 2
Time Frame: Baseline to Day 2
Reporting Status: Not Posted

3. Secondary Outcome: Mean Change in Intraocular Pressure at Day 3
Time Frame: Baseline to Day 3
Reporting Status: Not Posted

4. Secondary Outcome: Mean Change in Intraocular Pressure at Day 4
Time Frame: Baseline to Day 4
Reporting Status: Not Posted

5. Secondary Outcome: Mean Change in Intraocular Pressure at Day 5
Time Frame: Day 4 to Day 5
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | High Dose Drug Device/ Bimatoprost 0.03% | Low Dose Drug Device / Bimatoprost 0.03% | Placebo Device / Bimatoprost 0.03%
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/12 | 0/18
Other Adverse Events (participants affected / at risk) | 12/17 | 7/12 | 8/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | High Dose Drug Device/ Bimatoprost 0.03% (N=17) | Low Dose Drug Device / Bimatoprost 0.03% (N=12) | Placebo Device / Bimatoprost 0.03% (N=18)
Conjunctival Hyperemia (Eye disorders) | 5 (5) | 4 (4) | 5 (5)
Eye Irritation (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Eye Pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye Pruritus (Eye disorders) | 2 (2) | 1 (1) | 0 (0)
Eyelid Pruritus (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Eyelid Margin Crusting (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eyelid Oedema (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Foreign Body Sensation in Eye (Eye disorders) | 1 (1) | 1 (2) | 0 (0)
Punctate Keratitis (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Ocular Hyperemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Lid Margin Discharge (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abnormal Sensation in Eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye Disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Medical Device Complication (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 3 (3)
Medical Device Discomfort (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0/0 (0) | 2 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication requires written consent of the sponsor.